CLINICAL TRIAL: NCT05894005
Title: The Efficacy of Immersive 360-degree Video in Improving Spatial Orientation Among Medical Students.
Brief Title: The Use of Immersive 360-degree Video in Improving Spatial Orientation
Acronym: IMProVe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 5856
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Virtual Reality
Keywords: Education, Virtual Reality, Orientation
MeSH Terms: conditions — Orientation, Spatial

STUDY DESIGN:
Intervention Model Description: Participants will be asked to complete a navigation task within Sunnybrook Hospital. Prior to the task, video instructions will be provided using either 2D video or immersive 360-degree VR video.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not be aware of which video format will be viewed by the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Immersive Virtual Reality (IVR)
  Interventions: Other: Immersive Virtual Reality (IVR)
- Group B (Active Comparator): Traditional 2-D Video
  Interventions: Other: Traditional 2-D Video

INTERVENTIONS:
Other: Immersive Virtual Reality (IVR) — Students will be first taken to the anesthesia lounge. Here the students will receive IVR instructions on how to navigate the route (i.e. they will watch a 360-degree video using Oculus VR headset). Then the students will be assessed with an observed walkthrough of the route.
  Arms: Group A
Other: Traditional 2-D Video — Students will be first taken to the anesthesia lounge. Students will receive 2D video instruction on how to navigate the route by watching a normal 2D video using a desktop computer screen. Then the students will be assessed with an observed walkthrough of the route.
  Arms: Group B

SUMMARY:
As medical students rotate through different hospital sites as part of their studies, the students are frequently exposed to new and unfamiliar environments. This can cause anxiety in some students, and can potentially result in students becoming lost, and arriving late to their activities. To prevent this, students are currently provided with instructions in the form of written directions, photographs, maps, and/or 2-dimensional videos.

In this study, the investigators will test if immersive 360-degree virtual reality videos (videos shown using a headset/goggles that allow the wearer to experience the video as though they were actually there), are better at teaching medical students how to navigate the hospital and find new locations, compared to normal, 2-dimensional video instructions.

Medical students will be asked to find their way to a new location within the hospital, after being given instructions using either 2-dimensional (standard) video or 360-degree virtual reality video. The investigators will measure how long it takes students to find the new location, and how often the students get lost or confused along the way.

If successful, the investigators believe that this new method of teaching will help students to get around in new places more easily and lessen student anxiety. This will also increase knowledge related to 360-degree virtual reality video for teaching medical students.

DETAILED DESCRIPTION:
Background and Rationale: Effective medical education requires continuous adaptation, including adoption of new technologies. Readily affordable and accessible new technologies have the potential to improve trainee performance, build their confidence, and prepare them for the demands of clinical care. At their best, new medical education technologies achieve these goals without requiring a significant investment of time and resources, which are understandably limited in the modern education system. A classic example is the adoption of 2-dimensional (2D) videos for medical training, which can provide a standardized and consistent learning experience that enhances knowledge transfer, appeals to learners with various learning styles, and allows for both synchronous and asynchronous teaching.

An emerging and promising technology for use in medical education is immersive virtual reality (IVR). Combined with a head-mounted display (such as a VR headset), this technology fully immerses the user in a virtual setting, allowing the user to feel present in the virtual space. As commercial VR headsets become readily affordable and available, IVR presents as a cost-effective educational tool that does not require significant time and resources such as staff and hospital spaces.

There is a growing literature on the use of IVR in medical education. A recent systematic review found that trainees were very receptive to IVR, rating it more highly than most other training methods. Users found IVR to be a "positive learning experience, increasing self-efficacy, attentiveness, and motivation". Furthermore, IVR can be highly effective: when compared with other training methods, those trained with IVR had better performance scores for surgical procedures such as total hip arthroplasty or tibia intramedullary nailing. However, it must be noted that IVR is not universally superior to other training methods. For instance, IVR was similar to existing study materials for learning medical knowledge about total hip arthroplasty and anatomy, or general lower cognitive skills such as remembering facts. Thus, IVR must be tested on a case-by-case basis before being adopted for a new medical education area.

One intriguing use for IVR is during onboarding and orientation of medical students. Throughout their training, undergraduate medical students rotate through different clinical sites, where they often face the challenge of adjusting to unfamiliar environments. This unfamiliarity may cause students to get lost and arrive late to their clinical assignments. This is a known issue: a survey of surgical clerkship students at a US hospital found that over 30% of respondents wanted more tours of the hospital early in their clerkship. Anecdotal and survey feedback from Sunnybrook Health Sciences Centre also suggests that unfamiliarity with a new environment induces anxiety among trainees and may result in some 'false' starts on the first day of the rotations. Given that stress and anxiety is associated with impaired medical student learning and burnout, strategies that improve wayfinding for medical students will positively impact their learning, confidence, and overall education experience.

Currently, wayfinding and orientation for medical students primarily utilize text-based directions, which are at times supplemented by photographs and standard 2D videos. The addition of such 2D videos for hospital induction has been shown to improve learners' experiences, allowing them to feel more confident and better oriented on the first day of their placement. Compared to 2D videos, the realism of IVR utilizing 360-degree immersive videos may provide a sense of direction with better wayfinding skills, because it will allow the learner to explore and experience the depicted location. This notion is supported by a 2017 systematic review, which found IVR to be particularly effective in improving users' spatial learning and orientation. However, whether 360-degree video IVR is superior to 2D videos on improving the wayfinding and orientation experience for medical students has not been studied in a randomized trial.

The goal of this study is to evaluate the effectiveness of 360-degree video IVR in preparing medical students to enhance both wayfinding and their subjective experience in an unfamiliar hospital environment.

Objectives

Primary objective: To determine whether 360-degree video IVR enhances spatial orientation for pre-clerkship students compared to 2D video. The investigators will measure the time, distance travelled, and error rate of learners as they travel to their destinations.

Secondary objective: To determine whether 360-degree video IVR enhances student confidence and reduces their anxiety compared to 2D video. Questionnaires will assess learners' subjective experience with IVR and 2D video orientation.

Study design and recruitment: The proposed study is a single-center, prospective, balanced (1:1) randomized, assessor-blinded, parallel group design-controlled trial. Pre-clerkship (year 1 and 2) medical students from the University of Toronto, Faculty of Medicine will be invited to take part in the study using a recruitment email. The exclusion criteria are prior experience visiting Sunnybrook Health Sciences Centre for personal reasons or previous coursework, shadowing, research, or clinical rotations.

Methodology: Each student-participant will be required to complete one route at Sunnybrook Hospital: from the anesthesia lounge on the 3rd floor to the fracture clinic (CG 15) on the ground floor using the B wing stairs.

The Under Armour® smartphone application (https://www.mapmyrun.com) was used to ensure the distance of the route (approximately 100 m), which would take approximately two minutes to walk.

Prior to completing the route, students will receive 360-degree video IVR or 2D video instruction on navigating the route. One group of participants will receive IVR instruction for the route. The other group will receive 2D video instruction for the route.

Randomization:

A computer-generated random number sequence has been generated using the Sealed Envelope online randomization database (https://www.sealedenvelope.com) and used to allocate participants 1:1 to Group A or B (described below). Randomization will take place on the day of the study, using sequentially numbered opaque envelopes.

Study Groups

* Group A IVR: Students will be first taken to the anesthesia lounge. Here the students will receive IVR instructions on how to navigate the route (i.e. they will watch a 360-degree video using Oculus VR headset). Then the students will be assessed with an observed walkthrough of the route
* Group B 2D video: Students will be first taken to the anesthesia lounge. Students will receive 2D video instruction on how to navigate the route by watching a normal 2D video using a desktop computer screen. Then the students will be assessed with an observed walkthrough of the route.

Work Plan:

On the day of the study, participants will complete a baseline questionnaire collecting data on key potentially confounding factors such as previous IVR experience, self-described navigation ability, and formal navigation training.

Following randomization, participants will be allowed to watch the video (360-degree or 2D) once but can repeat watch if they feel that they missed something on their first watch. There will be a 5-minute cool off period after the video and before the navigation task is attempted. A blinded observer will accompany the participant on their route and time their performance, as well as count any wayfinding errors and corrective measures.

Participants' confidence and anxiety will be assessed before and after receiving 2D/IVR instructions. After completing the route, participants will be asked to rate the extent to which the instructions helped them navigate the hospital and reduce their anxiety and complete a questionnaire on their comfort and satisfaction with IVR or 2D video instruction.

Sample size:

If the Route 2-D video participants take approximately 148 ± 38 seconds (based on an exploratory phase of the study) to complete the route, the investigators aim to demonstrate that the Route 3-D IVR participants can complete the route within 110 ± 38 seconds. Using conventional measures, with a Type I error rate of 0.05 and a Type II error rate of 0.1 (i.e., 90% power), the investigators estimate that they will need 44 participants, with 22 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Pre-clerkship (year 1 and 2) medical students from the University of Toronto, Temerty Faculty of Medicine.

Exclusion Criteria:

* Experience visiting Sunnybrook for personal reasons or previous coursework, shadowing, research, or clinical rotations. Having a familiarity with the floor plan of the hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-11-08 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Time assessment | 1 hour
  A blinded research assistant will follow and time how long it takes the medical student to travel from the starting to end point.

SECONDARY OUTCOMES:
Distance assessment: | 1 hour
  The number of steps and distance travelled will be measured using a standardized pedometer
Way-finding corrective measures: | 1 hour
  1. Number of wrong turns/wrong floors/doors entered 2. Number of times student asks for help.
Satisfaction Survey | 1 hour
  Comfort and satisfaction in learning through VR and traditional methods.

CONTACTS AND LOCATIONS:
Overall Officials: Ahtsham U Niazi, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abraham R, Adiga I, George B. Orienting incoming medical students to the process of PBL through video. Educ Health (Abingdon). 2011 Aug;24(2):582. Epub 2011 Aug 2. No abstract available. PMID 22081660
- [Background] Alaker M, Wynn GR, Arulampalam T. Virtual reality training in laparoscopic surgery: A systematic review & meta-analysis. Int J Surg. 2016 May;29:85-94. doi: 10.1016/j.ijsu.2016.03.034. Epub 2016 Mar 15. PMID 26992652
- [Background] Barsom EZ, Graafland M, Schijven MP. Systematic review on the effectiveness of augmented reality applications in medical training. Surg Endosc. 2016 Oct;30(10):4174-83. doi: 10.1007/s00464-016-4800-6. Epub 2016 Feb 23. PMID 26905573
- [Background] Bridge PD, Jackson M, Robinson L. The effectiveness of streaming video on medical student learning: a case study. Med Educ Online. 2009 Aug 19;14:11. doi: 10.3885/meo.2009.Res00311. PMID 20165525
- [Background] Cha YW, Dou M, Chabra R, Menozzi F, State A, Wallen E, Fuchs H. Immersive Learning Experiences for Surgical Procedures. Stud Health Technol Inform. 2016;220:55-62. PMID 27046554
- [Background] de Leng B, Dolmans D, van de Wiel M, Muijtjens A, van der Vleuten C. How video cases should be used as authentic stimuli in problem-based medical education. Med Educ. 2007 Feb;41(2):181-8. doi: 10.1111/j.1365-2929.2006.02671.x. PMID 17269952
- [Background] Flores AS, Garber SM, Niesen AD, Long TR, Lynch JJ, Wass CT. Clinical application of a novel video camera laryngoscope: a case series venturing beyond the normal airway. J Clin Anesth. 2010 May;22(3):201-4. doi: 10.1016/j.jclinane.2009.03.016. PMID 20400007
- [Background] Gagliano ME. A literature review on the efficacy of video in patient education. J Med Educ. 1988 Oct;63(10):785-92. doi: 10.1097/00001888-198810000-00006. PMID 3050102
- [Background] Gandsas A, McIntire K, Palli G, Park A. Live streaming video for medical education: a laboratory model. J Laparoendosc Adv Surg Tech A. 2002 Oct;12(5):377-82. doi: 10.1089/109264202320884135. PMID 12470413
- [Background] Knowles C, Kinchington F, Erwin J, Peters B. A randomised controlled trial of the effectiveness of combining video role play with traditional methods of delivering undergraduate medical education. Sex Transm Infect. 2001 Oct;77(5):376-80. doi: 10.1136/sti.77.5.376. PMID 11588286
- [Background] Spofford CM, Bayman EO, Szeluga DJ, From RP. Anesthesia machine checkout and room setup: a randomized, single-blind, comparison of two teaching modalities. J Educ Perioper Med. 2012 Jan 1;14(1):E060. eCollection 2012 Jan-Jun. PMID 27175391
- [Background] Zhu E, Hadadgar A, Masiello I, Zary N. Augmented reality in healthcare education: an integrative review. PeerJ. 2014 Jul 8;2:e469. doi: 10.7717/peerj.469. eCollection 2014. PMID 25071992